CLINICAL TRIAL: NCT00928850
Title: A Randomized Trial of Modifications to Radical Prostatectomy: Feasibility Study
Brief Title: Modifications to Radical Prostatectomy: Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-051
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Prostate Cancer
Keywords: Prostate; Radical Prostatectomy; urethral irrigation; fascial suturing; 09-051
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (4):
- urethral irrigation but no fascial suturing, QOL forms (Active Comparator): The anterior two-thirds of the urethra is divided exposing a Foley catheter that was placed at the beginning of the procedure. Irrigation of the urethra may prevent spread of prostate cancer cells to tissue that is not removed during surgery. The urethra is irrigated with 60 cc of sterile water as it is withdrawn from the patient to 'wash' the urethra.
  Interventions: Procedure: radical prostatectomy with urethral irrigation but no fascial suturing, QOL forms
- fascial suturing but no urethral irrigation, QOL forms (Active Comparator): For patients undergoing fascial suturing only, after the initial placement of the suture through the urethra a second bite is taken deeply into the fascia of the lateral pelvic fascia.
  Interventions: Procedure: radical prostatectomy with fascial suturing but no urethral irrigation, QOL forms
- both urethral irrigation and fascial suturing, QOL forms (Active Comparator)
  Interventions: Procedure: radical prostatectomy with both urethral irrigation and fascial suturing, QOL forms
- neither urethral irrigation nor fascial suturing, QOL forms (Active Comparator)
  Interventions: Procedure: radical prostatectomy with neither urethral irrigation nor fascial suturing, QOL forms

INTERVENTIONS:
Procedure: radical prostatectomy with urethral irrigation but no fascial suturing, QOL forms — Cancer cells can spill during surgery and this can cause cancer to return ("recur"). Some surgeons believe that "irrigating" could help stop spilling of cancer cells. "Irrigating" means washing the surgical area with sterile water and sucking the water back up through a tube. As a result, surgeons vary as to how they irrigate. In this study, we will examine irrigation of the urethra. This is the part of the body that carries urine from the bladder to the penis. Quality of life are assessed for clinical evaluation approximately 3, 6, 9, 12, 18, 24, 36 and 48 months after surgery
  Arms: urethral irrigation but no fascial suturing, QOL forms
Procedure: radical prostatectomy with fascial suturing but no urethral irrigation, QOL forms — Surgeons believe that what happens to the urethra can affect the risk of incontinence. This is when a patient cannot control urine, and drips or leaks urine. One idea is that additional stitches ("sutures") to the connective tissue ("fascia") could be helpful, but this is not known for sure. Quality of life are assessed for clinical evaluation approximately 3, 6, 9, 12, 18, 24, 36 and 48 months after surgery
  Arms: fascial suturing but no urethral irrigation, QOL forms
Procedure: radical prostatectomy with both urethral irrigation and fascial suturing, QOL forms — Quality of life are assessed for clinical evaluation approximately 3, 6, 9, 12, 18, 24, 36 and 48 months after surgery
  Arms: both urethral irrigation and fascial suturing, QOL forms
Procedure: radical prostatectomy with neither urethral irrigation nor fascial suturing, QOL forms — Quality of life are assessed for clinical evaluation approximately 3, 6, 9, 12, 18, 24, 36 and 48 months after surgery
  Arms: neither urethral irrigation nor fascial suturing, QOL forms

SUMMARY:
This study aims to determine whether surgeons at Memorial Sloan-Kettering Cancer Center are able to randomize patients to test modifications of surgery to remove the prostate. Surgery to remove the prostate is known as a "radical prostatectomy". Surgeons know many things about the best way to do a radical prostatectomy. However, there is disagreement about some aspects of surgery. Two modifications of surgery to remove the prostate (radical prostatectomy) identified for this study include Irrigation, and Fascial Suturing.

Two aspects of the operation may vary, fascial suturing and urethral irrigation. For each aspect, surgeons will use their clinical judgment as to the best interests of the patient. In other words, if there are clear reasons to use or avoid a fascial suturing approach, the surgeon will act accordingly; similarly, if there is a clear reason to irrigate or avoid irrigating the urethra, the surgeon can make the appropriate clinical decision. If the surgeon is unsure as to which approach to take, then the randomization scheme will be followed.

All of the surgeons who are taking part in this study have used these techniques at different times. However, they are unsure as to the best approach. Sometimes, they use different treatments with different patients.

Irrigation. Cancer cells can spill during surgery and this can cause cancer to return ("recur"). Some surgeons believe that "irrigating" could help stop spilling of cancer cells. "Irrigating" means washing the surgical area with sterile water and sucking the water back up through a tube. As a result, surgeons vary as to how they irrigate. In this study, we will examine irrigation of the urethra. This is the part of the body that carries urine from the bladder to the penis.

Fascial suturing. Surgeons believe that what happens to the urethra can affect the risk of incontinence. This is when a patient cannot control urine, and drips or leaks urine. One idea is that additional stitches ("sutures") to the connective tissue ("fascia") could be helpful, but this is not known for sure.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for radical prostatectomy for the treatment of prostate cancer with one of the consenting surgeons at MSKCC.

Exclusion Criteria:

* Prior treatment for prostate cancer: radiation, hormonal therapy, chemotherapy or focal therapy.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2009-06; Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
To pilot a randomized trial of modifications to radical prostatectomy to determine:Proportion of patients accrued and Accrual rate | 1 year

SECONDARY OUTCOMES:
Determine surgeon compliance with allocation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Vickers, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Vickers AJ, Bennette C, Touijer K, Coleman J, Laudone V, Carver B, Eastham JA, Scardino PT. Feasibility study of a clinically-integrated randomized trial of modifications to radical prostatectomy. Trials. 2012 Feb 24;13:23. doi: 10.1186/1745-6215-13-23. PMID 22364367
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org